CLINICAL TRIAL: NCT04474067
Title: A Multi-Center Study Evaluating Clinical Course in Patients With COVID-19 and Its Relationship to Cytokine Storm
Brief Title: COVID-19 - Cytokine Storm
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Barzilai Medical Center (Other); The Chaim Sheba Medical Center (Other)
Responsible Party: Principal Investigator, Mevorach Dror, Professor & Head, Department of Internal Medicine B; Head, Rheumatology Research Center, Hadassah and the Hebrew University Medical School, Hadassah Medical Organization
Other Study IDs: DM002
Record Dates: First submitted 2020-07-15; First posted 2020-07-16 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples obtained from patients with COVID-19, sepsis, or CAR T and cytokine storm following a consent, for a total amount of up to 10 ml of blood. Also, Blood leftover samples obtained from Hadassah biological blood bank, or from any routine blood examination, or a total amount of up to 10 ml of blood from hospitalized COVID-19 patients is retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- • Asymptomatic or Pre-symptomatic Infection: Individuals who test positive for SARS-CoV-2 by virologic testing using a molecular diagnostic (e.g., polymerase chain reaction) or antigen test, but have no symptoms.
  Interventions: Other: No intervention
- Mild COVID-19: Individuals who have any of the various signs and symptoms of COVID-19 (e.g., fever, cough, sore throat, malaise, headache, muscle pain) without shortness of breath, dyspnea, or abnormal chest imaging.
  According to NIH classification
  Interventions: Other: No intervention
- Moderate COVID-19: COVID-19 patients who have evidence of lower respiratory disease by clinical assessment or imaging and a saturation of oxygen (SpO2) ≥94% on room air at sea level.
  Interventions: Other: No intervention
- Severe COVID-19: COVID-19 patients who have respiratory frequency >30 breaths per minute, SpO2 <94% on room air at sea level, ratio of arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2) <300 mmHg, or lung infiltrates >50%
  Interventions: Other: No intervention
- Critical COVID-19: COVID-19 patients who have respiratory failure, septic shock, and/or multiple organ dysfunction.
  Interventions: Other: No intervention
- Sepsis: A control group of patients with sepsis-related cytokine storm
  Interventions: Other: No intervention
- CAR-T CRS: A control group of patients with cytokine release syndrome due to CAR-T therapy
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study, with no intervention.

SUMMARY:
This is a multi-center study comparing clinical outcomes in patients with COVID-19 in subjects hospitalized at Hadassah and other hospitals for PCR or serology confirmed COVID-19 and compare the outcomes to the presence of different degrees of a cytokine storm. The patients will be subdivided into a mild, moderate, and severe course according to NEWS2.

DETAILED DESCRIPTION:
Study Rationale

Over 100 patients were hospitalized at Hadassah in the recent 2 months with the diagnosis of COVID-19.

We would like to summarize the clinical outcomes and their correlation to a cytokine storm at Hadassah and additional hospitals and additional hospitals in Israel.

COVID-19, the name given to the clinical syndrome associated with the newly recognized virus SARS-CoV-2 has become pandemic with a mortality estimated based on reports from China between 1-3% and complications among hospitalized patients leading to up to 15-25% admissions to the ICU.

The clinical presentation includes both upper and lower respiratory tract infection, but patients may also be asymptomatic.

A diagnostic PCR assay was rapidly developed in Hong Kong and Berlin that accurately detects SARS-CoV-2 in samples from nose and throat swabs or sputum of hospitalized patients and is used by public-health authorities around the world.

To avoid cross-reactivity with SARS-CoV or other coronaviruses, the test detects a region of the gene encoding RNA-dependent RNA polymerase that is unique to SARS-CoV-2.

Not all patients need hospitalization but due to the high index of infection spread, all detected patients are put in isolation to prevent transmission of the infection to others.

The development of vaccines is undoubtedly an important step and several MERS vaccines were already in clinical trials when word of the new outbreak spread. However, developing and testing the correct viral protein that will be effective (and probably not 100% protective) will take some time.

In the meantime, anti-viral agents are tested including a combination of two human immunodeficiency virus (HIV) antivirals. Lopinavir and ritonavir have been taking center stage as potential therapies for COVID-19 and there are at least three registered randomized clinical trial testing the lopinavir-ritonavir combination in Chinese patients infected with SARS-CoV-2 (NCT04255017, NCT04252885 and NCT04251871) with the results of one being negative, as published in the New England Journal of Medicine in March 2020. A handful of other HIV antivirals are currently in clinical testing against SARS-CoV-2, including darunavir-cobicistat. , donated by the US pharmaceutical company Johnson & Johnson to the Shanghai Public Health Clinical Center. Nucleoside analogs are being considered too and Remdesivir was used to treat the first US patient infected with SARS-CoV-2, who recovered. It is also in phase 3 trials in Wuhan patients infected with SARS-CoV-2, overseen by the China-Japan Friendship Hospital in Beijing (NCT04252664 and NCT04257656). However, SARS-CoV-2 have its own proteases, including its main protease, Mpro, and HIV antivirals design are tailored specifically to block the activity of HIV proteases to avoid off-target effects on human cells, which makes them less likely to bind SARS-CoV-2 proteases as well. Chloroquine was recently suggested as an additional anti-viral medication. In addition, even if anti-viral therapy will be found to be efficacious against SARS-CoV-2, will this be the treatment of choice in patients admitted to the ICU? Not necessarily.

The term "cytokine storm" calls up vivid images of an immune system gone awry and an inflammatory response flaring out of control. The term has captured the attention of the public and the scientific community alike and is increasingly being used in both the popular media and the scientific literature. Indeed, a few publications have indicated an important part of the complications in COVID-19 are related to a cytokine storm (Huang et al. Lancet 2020, Mehta et al. Lancet 2020).

Taken together, in patients with moderate to severe COVID-19, there may be an underlying immunological mechanism of action that is a hyper-inflammatory pathway associated with increased death.

Study Design

A multi-center study comparing clinical outcomes in patients with COVID-19 in subjects hospitalized at Hadassah and other hospitals for PCR or serology confirmed COVID-19 and compare the outcomes to the presence of different degrees of a cytokine storm.

The patients will be subdivided into five severities of COVID-19 illness according to the new NIH Patient Classification (www.covid19treatmentguidelines.nih.gov/overview/management-of-covid-19/):

* Asymptomatic or Pre-symptomatic Infection: Individuals who test positive for SARS-CoV-2 by virologic testing using a molecular diagnostic (e.g., polymerase chain reaction) or antigen test, but have no symptoms.
* Mild Illness: Individuals who have any of the various signs and symptoms of COVID-19 (e.g., fever, cough, sore throat, malaise, headache, muscle pain) without shortness of breath, dyspnea, or abnormal chest imaging.
* Moderate Illness: Individuals who have evidence of lower respiratory disease by clinical assessment or imaging and a saturation of oxygen (SpO2) ≥94% on room air at sea level.
* Severe Illness: Individuals who have respiratory frequency >30 breaths per minute, SpO2 <94% on room air at sea level, ratio of arterial partial pressure of oxygen to fraction of inspired oxygen (PaO2/FiO2) <300 mmHg, or lung infiltrates >50%
* Critical Illness: Individuals who have respiratory failure, septic shock, and/or multiple organ dysfunction.

The cytokine storm will be compared to cytokine storm in sepsis and in chimeric antigen receptor (CAR)-T therapy, associated with Cytokine release Syndrome (CRS).

Handling of blood samples

Blood results will be taken from the Hospital clinical evaluation system (MAHAR). Blood leftover samples obtained from Hadassah biological blood bank, or for serological confirmation or IL6 level tests (as a rationale for injecting tocilizumab, or from any routine blood examination, will be used for cytokines/chemokines/hematopoietic growth factors/ Complement/ DNA methylation measurements.

In the case of hospitalized patients, a total amount of up to 10 ml of blood will be drawn. Blood samples will be obtained and handled according to the institutional guidelines and approvals.

Statistical Analysis

The data will be summarized by different clinical outcomes listing the mean, standard deviation, minimum, median, maximum, and number of subjects for continuous data, or in tables listing count and percentage for categorical and event data, as appropriate. Descriptive analyses and, where appropriate, statistical testing will compare between each of the subgroups.

All statistical analyses will be performed, and data appendixes will be created using the SAS® system (SAS Institute, Cary, NC), Version 9.4, or higher.

ELIGIBILITY:
Inclusion Criteria:

Patients, male or female of any age diagnosed with COVID-19, as defined below:

1. Laboratory confirmation of SARS-CoV-2 infection by reverse transcription-polymerase chain reaction (RT-PCR) from any diagnostic sampling source.

   OR
2. Serological evidence of SARS-CoV-2 infection

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients that were hospitalized at Hadassah Medical Center and other hospitals in Israel, with the diagnosis of COVID-19 (as specified in the inclusion criteria).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-06-28 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Clinical Outcomes of Patients with COVID-19 using the National Early Warning Score 2 (NEWS2) system | 6 months
  To compare the clinical outcomes of patients with COVID-19 to Sepsis and CAR-T-related cytokine storm.
  This will be done by assessment of acute-illness severity using the NEWS2 scoring system (Higher scores mean more severe illness)
Clinical Outcomes of Patients with COVID-19 using the new NIH Patient Classification of severity of illness | 6 months
  To compare the clinical outcomes of patients with COVID-19 to Sepsis and CAR-T-related cytokine storm.
  This will be done by assessment of acute-illness severity using the new NIH Patient Classification to (1) Asymptomatic or Pre-symptomatic Infection; (2) Mild Illness; (3) Moderate Illness; (4) Severe Illness; (5) Critical Illness As detailed in the Study design section.
Mortality | 6 months
  Incidence rate of Mortality from any cause
Cytokine/Chemokine/Hematopoietic Growth Factors/ Complement and Other Immune Modulators in Patients with COVID-19 | 6 months
  To assess cytokine/chemokine/hematopoietic growth factors/ Complement and other immune modulators in patients with COVID-19 by measuring the serum concentrations of these factors in COVID-19 patients and compare those the levels of patients with sepsis and CAR T cytokine release syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Dror Mevorach, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Siddiqi HK, Mehra MR. COVID-19 illness in native and immunosuppressed states: A clinical-therapeutic staging proposal. J Heart Lung Transplant. 2020 May;39(5):405-407. doi: 10.1016/j.healun.2020.03.012. Epub 2020 Mar 20. No abstract available. PMID 32362390
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578